CLINICAL TRIAL: NCT02107066
Title: Impact of Exercise on Ovarian Cancer Prognosis
Brief Title: Women's Activity and Lifestyle Study in Connecticut
Acronym: WALC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0904004976; R01CA138556 (NIH)
Record Dates: First submitted 2012-05-17; First posted 2014-04-08 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2014-04

CONDITIONS: Ovarian Cancer
Keywords: exercise; physical activity; ovarian cancer; quality of life; fatigue; weight
MeSH Terms: conditions — Ovarian Neoplasms; Motor Activity; Fatigue; Body Weight | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- attention control (Active Comparator): Women randomized to attention control will receive the same attention as women randomized to exercise intervention, i.e., weekly phone calls for 6 months. Each call is about 15 min. Women in the attention control will receive information on ovarian cancer health education topics.
  Interventions: Behavioral: Exercise
- exercise (Experimental): Women randomized to exercise will receive telephone-counseling weekly for 6 months to increase their exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Weekly telephone counseling to increase aerobic exercise to 150 min/wk for 6 months.

SUMMARY:
Despite an increase in longevity, surviving ovarian cancer often brings an array of unpleasant side effects and compromises in QOL. Our proposed trial will be the first study to test whether exercise compared with attention control has a beneficial impact on quality of life, fitness and surrogate markers of ovarian cancer. Our trial could suggest a unique and important role for exercise in ovarian cancer care given that physical and functional aspects of QOL are often the most compromised in ovarian cancer patients.

DETAILED DESCRIPTION:
Currently, the American Cancer Society recommends a physically active lifestyle for cancer survivors to increase disease-free survival from cancer and other chronic diseases, and to improve quality of life. Studies of a strong benefit of physical activity on improving QOL following other types of cancer treatment, e.g., breast cancer, are well documented in the literature; yet very few studies of physical activity and QOL after a diagnosis of ovarian cancer have been published. Therefore, clinical trials of exercise on common physical and psychological consequences of ovarian cancer and its treatments are warranted.

The primary aims of our study are to examine, in 230 women who have completed treatment for Stage I-IV ovarian cancer, the impact of a moderate-intensity aerobic exercise intervention vs. attention control on:

* Quality of Life
* Body Composition (weight, BMI, total and % body fat, waist and hip circumference)
* Hormones possibly associated with physical activity and ovarian cancer prognosis (insulin, IGF-I, IGF-II, IGF binding protein-3, CRP, leptin, estrone, estradiol, free estradiol, and sex-hormone binding globulin, osteopontin, MIF, prolactin, and CA-125)
* Cardiorespiratory Fitness - an objective measure of functional capacity and adherence to exercise.

Hypotheses: Women randomized to exercise will experience improvements in quality of life, body composition, hormone levels, and cardiorespiratory fitness compared to women randomized to usual care.

Our trial could suggest a unique and important role for exercise in ovarian cancer care given that physical and functional aspects of QOL are often the most compromised in ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* stage I-IV ovarian cancer
* less than 76 yrs of age

Exclusion Criteria:

* exercising

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Functional Assessment of Cancer Therapy-Ovarian (FACT-O) | 6 months
  The FACT-General (FACT-G) consists of four subscales that measure wellbeing in physical, social, emotional and functional domains. The FACT-Ovarian (FACT-O) is a disease-specific measure and is comprised of the four subscales from the FACT-G in addition to a set of items that address concerns specific to ovarian cancer
Change from Baseline in Functional Assessment of Cancer Therapy-Fatigue (FACT-F) | 6 months
  FACT-F is a self-reporting questionnaire comprised of 13 fatigue-related items. Each item on the FACT-F is answered on a five-point scale and summed, with total scores ranging between 0 and 52. Lower scores indicate greater self-reported fatigue.
Change from Baseline in Short Form 36 (SF-36) | 6 months
  The SF-36 survey was interpreted using eight subscales (emotional, functional, pain, physical, roles-emotional, roles-physical, social, vitality) that can be combined into physical (PCS) and mental (MCS) component summary scores. The PCS score describes physical health and is composed of the general health, pain, physical functioning, and role-physical subscales. The MCS score describes mental health and is comprised of mental health, role-emotional, social functioning, and vitality subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Irwin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Cao A, Cartmel B, Li FY, Gottlieb LT, Harrigan M, Ligibel JA, Gogoi R, Schwartz PE, Esserman DA, Irwin ML, Ferrucci LM. Effect of Exercise on Chemotherapy-Induced Peripheral Neuropathy Among Patients Treated for Ovarian Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2326463. doi: 10.1001/jamanetworkopen.2023.26463. PMID 37526937
- [Derived] Cartmel B, Li FY, Zhou Y, Gottlieb L, Lu L, Mszar R, Harrigan M, Ligibel JA, Gogoi R, Schwartz PE, Risch HA, Irwin ML. Randomized trial of exercise on cancer-related blood biomarkers and survival in women with ovarian cancer. Cancer Med. 2023 Jul;12(14):15492-15503. doi: 10.1002/cam4.6187. Epub 2023 Jun 3. PMID 37269192
- [Derived] Cao A, Cartmel B, Li FY, Gottlieb LT, Harrigan M, Ligibel JA, Gogoi R, Schwartz PE, Irwin ML, Ferrucci LM. Effect of exercise on body composition among women with ovarian cancer. J Cancer Surviv. 2023 Oct;17(5):1386-1396. doi: 10.1007/s11764-022-01207-x. Epub 2022 Apr 4. PMID 35377104